CLINICAL TRIAL: NCT04543981
Title: Prevalence of the Signs and Symptoms of Tempro-mandibular Joint Disorder in a Sample of Egyptian Adolescents According to Diagnostic Criteria for Tempro-mandibular Disorders(DC/TMD):A Cross Sectional Study
Brief Title: Prevalence of the Signs and Symptoms of TMD in Adolescents
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelrahman Abdelaleem, Master dgree student, Cairo University
Other Study IDs: ORTH 1-1-1
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: TMJ Disorder; TMD
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic Criteria for Tempro-mandibular Disorders(DC/TMD) — diagnostic sheet include questions to be answered by the patients and others include examinations will be done by the investigator

SUMMARY:
the Prevalence of the Signs and Symptoms of Tempro-mandibular Joint Disorder in a sample of Egyptian adolescents

DETAILED DESCRIPTION:
Our study is observational cross sectional study to evaluate the prevalence ofTempro-mandibular Joint Disorder( TMDs) in Egyptian adolescents based on Diagnostic Criteria for Tempro-mandibular Disorders(DC/TMD) .The following examinationwill be done for each patient and recorded in his/her chart:

Include maximal mandibular opening capacity, joint noises, deviation of mandible during opening and closing, tenderness of the TMJ and masticatory muscles, headache and pain in TMJ area.

All clinical examinations will be carried out by one investigator. Examination of TMJ disorders include the following aspects: I) Examination of TMJ sounds (clicking and crepitus) using a stethoscope over the TMJ area and by having the patient open and close the mouth.

II) Associated muscle disorders will be determined by:

1. palpation of TMJ area.
2. digital palpation and functional manipulation of the masticatory muscles according to Okeson.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents(age range10-18 years old).
* A well-defined dentalCl I, Cl II/1, Cl II/2, and Cl III relationship (Angle Classification).
* Mixed and permanent dentition.
* Both sexes.
* Normal skeletal pattern

Exclusion Criteria:

* Adolescents with syndromes.
* Systemic diseases affecting bones.
* Adolescents with rheumatoid arthritis.
* Previous trauma in the face.
* Neurological disorders.
* Psychiatric disorders.
* Neoplasia.
* Adolescents who had received orthodontic treatment.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: DC/TMD shhts will be assessed and obtained from adolescents in Diagnostic center clinic at the faculty of Dentistry, Cairo University
Sampling Method: Non-Probability Sample
Enrollment: 733 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
TMD | at the time of examination of each participant
  adolescents diagnosed positively for any TMD subtype (overall TMD) by DC/TMD.

SECONDARY OUTCOMES:
Myofacial pain | at the time of examination of each participant
  pain in each muscle of mastication will be recorded
mouth opening | at the time of examination of each participant
  limitation of mouth opening and pain during such movement
TMJ noises | at the time of examination of each participant
  Clicking and crepitus in tempro-mandibular joint

CONTACTS AND LOCATIONS:
Overall Officials: Manal foda, professor, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Cairo/Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided